CLINICAL TRIAL: NCT00619034
Title: Pharmacological Intervention Against Diabetic Retinal Flow Disturbances.
Brief Title: Pharmacological Intervention in Diabetic Retinopathy
Acronym: XAVOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Øjenafd. J, Department of Ophthalmology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2007-001697-84; XAVOT
Record Dates: First submitted 2008-02-07; First posted 2008-02-20 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-12

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Latanoprost; Diclofenac; dorzolamide; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- latanoprost (Experimental): Medical intervention cross-over
  Interventions: Drug: Latanoprost, diclofenac and dorzolamide (eyedrops)
- diclofenac (Active Comparator): medical intervention
  Interventions: Drug: Diclofenac
- dorzolamide (Experimental): dorzolamide eyedrops twice daily in one week
  Interventions: Drug: Dorzolamide

INTERVENTIONS:
Drug: Latanoprost, diclofenac and dorzolamide (eyedrops) — 1 eyedrop twice daily in one week
  Other Names: Xalatan; Voltaren ophtha; Trusopt
  Arms: latanoprost
Drug: Diclofenac — dicolfenac eyedrops twice daily i one eye
  Other Names: Voltaren ophtha
  Arms: diclofenac
Drug: Dorzolamide — dorzolamide eyedrops twice daily, in one eye for one week
  Other Names: Trusopt eyedrops
  Arms: dorzolamide

SUMMARY:
The purpose of this study is to determine if diabetic retinopathy can be treated with prostaglandin analogues, prostaglandin synthesis inhibitors or carbonic anhydrases inhibitors.

DETAILED DESCRIPTION:
Disturbances in retinal perfusion is believed to be involved in the pathophysiology of diabetic retinopathy. These disturbances may be due to changes in the basal diameter of retinal arterioles and to disturbances in the autoregulation of the diameter of these vessels when the blood pressure and the retinal metabolism changes. In vitro studies have shown that prostaglandins and carbonic anhydrases inhibitors are involved in the tone regulation of retinal arterioles, but it is unknown whether this finding is relevant in clinical practice. This can be tested in vivo by an retinal vessel analyzer measuring the dynamics of the retinal vessel diameter changes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 1 with moderate diabetic retinopathy/healthy
* Blood pressure < 135/85 mmHg

Exclusion Criteria:

* Eye disease (excluding diabetic retinopathy)
* Allergic
* Kidney disease
* Liver disease
* Severe asthma
* Heart disease
* Hypertension arterial
* Users of drugs that influence the metabolism of the prostaglandins in the carbon dioxide
* Pregnant and breastfeeding women and women who don't use secure contraception
* Persons who can't do without contact lens in the treated eye.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Diameter of retinal blood vessels | one year

SECONDARY OUTCOMES:
Influence on retinal blood flow in diabetes | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kathrine K Tilma, MD, Principal Investigator — Department of Ophthalmology - Aarhus, Denmark
Locations (1):
- Department of Ophthalmology, Aarhus, Denmark